CLINICAL TRIAL: NCT02462629
Title: A Phase 1 Dose-escalation and Expansion Study of BLZ-100 in Pediatric Subjects With Primary Central Nervous System Tumors
Brief Title: Study of BLZ-100 in Pediatric Subjects With CNS Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blaze Bioscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BB-004
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Central Nervous System Tumors
Keywords: central nervous system tumor; BLZ-100; pediatrics; Tumor Paint; brain cancer; tozuleristide
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — tozuleristide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BLZ-100 (Experimental)
  Interventions: Drug: BLZ-100

INTERVENTIONS:
Drug: BLZ-100
  Other Names: Tumor Paint; tozuleristide

SUMMARY:
Many types of cancer are primarily treated with surgery and patient survival is directly related to the extent to which the tumor is able to be removed. It is often difficult for surgeons to distinguish tumor tissue from normal tissue or to detect tumor cells that have spread from the original tumor site, resulting in incomplete removal of the tumor and reduced patient survival. In some sites, such as the brain, it is critical to avoid damage to normal tissue around the tumor to prevent adverse effects of surgery on function. The investigators hypothesize that BLZ-100 will improve surgical outcomes by allowing surgeons to visualize the edges of the tumor and small groups of cancer cells that have spread to other sites in real-time as they operate. This is a safety study to assess the safety of BLZ-100 in pediatric patients with central nervous system tumors.

DETAILED DESCRIPTION:
Subjects who provide voluntary written informed consent, or have it provided by their legally acceptable representative, will be screened for eligibility. Subjects meeting all of the inclusion and none of the exclusion criteria will be eligible to participate.

Subjects will be required to arrive at the hospital for dosing at least 1 hour before the planned surgical excision. Following dosing, subjects will be monitored for safety and surgical excision will occur at least 1 hour after study product administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age: >1 month and <30 years at time of enrollment
2. Diagnosis: Must have MRI documenting a measurable lesion w/in central nervous system consistent with primary central nervous system tumor, for which maximal safe surgical resection is indicated
3. Timing of surgery: Must be anticipated to take place at least 1 hour after BLZ-100 administration
4. Prior therapy: Must have recovered from acute toxic effects of prior anti-cancer therapy (durations relative to date of enrollment):

   * Radiation therapy: may not have had radiation therapy to area of tumor planned to be resected w/in 28 days
   * Chemotherapy: ≥14 days from any myelosuppressive chemotherapy and abs neutrophil ct ≥1000/mm3 , 42 days if prior nitrosurea
   * Biologic: ≥7 days from anti-neoplastic biologic agent
   * Immunotherapy: ≥42 days after completion of immunotherapy
   * Monoclonal antibody: ≥3 half-lives of antibody since last admin.
5. Organ function requirements:

   * Adequate renal function defined as:

     * serum creatinine w/in normal limits or
     * calculated creatinine clearance > 100 mL/min/1.73 m2
   * Adequate liver function defined as:

     * bilirubin <2x upper limit of normal for age
     * alanine aminotransferase <3x upper limit of normal for age (<135 U/mL)
     * serum albumin >2g/dL
   * Adequate coagulation defined as:

     * no evidence of active/clinically significant bleeding. May be evidence of punctate hemorrhage w/in tumor as long as not considered clinically significant to warrant urgent surgical evacuation
     * internal normalized ratio and partial thromboplastin time <1.5x upper limit of normal
6. Informed Consent: Written informed consent must be obtained from subject or parent/legal guardian prior to enrollment. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

1. Pregnancy and contraception: Subjects who are pregnant, breast-feeding or planning to conceive within 30 days are not eligible
2. Concomitant medications:

   * Corticosteroids: no restrictions
   * Investigational drugs: must not be receiving other investigational (from other studies) drugs at time of enrollment and must not be planning to take other investigational drugs during DLT period
   * Anti-cancer agents: must not be receiving other anti-cancer agents at time of enrollment and must not be planning to take other anti-cancer agents during DLT period
   * Anticoagulation: if currently receiving therapeutic anticoagulation with heparin, low-molecular weight heparin, or Coumadin, not eligible
   * Anti-platelet agents: if currently receiving aspirin, ibuprofen or other non-steroidal anti-inflammatory or anti-platelet agents, not eligible
   * Photosensitizing drugs, medications which might generate fluorescence or according to label, might generate photochemical reaction. These include hematoporphyrin derivatives and purified fractions; Photofrin®; and precursors of protoporphyrin IX (5-Aminolevulinic acid) used in Gliolan or Hexvix
   * Subjects must not have received BLZ-100 within 30 days prior to re-treatment
3. Infection: Subjects with uncontrolled infection not eligible
4. Bleeding and Thrombosis:

   * If active bleeding requiring acute surgical intervention, not eligible
   * Subjects with stroke, arterial or venous thrombosis within 6 months not eligible
   * Subjects requiring anticoagulation not eligible
5. Acuity of surgical needs: Subjects with acute neurologic compromise, symptoms of impending cerebral herniation, or other condition(s) necessitating urgent or emergent neurosurgical intervention to be planned within 2 hours not eligible. NOTE: If subject is enrolled on study, receives study medication and subsequently condition worsens such that urgent surgical intervention is felt to be in best interest of subject, best interest of subject should always take precedence over timing between study medication and surgery
6. Required observations: Subjects who in opinion of investigator may not be able to comply with required safety and monitoring requirements are not eligible

Ages: 1 Month to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Seven days after study drug administration
  Safety will be assessed by physical examination and measurement of vital signs and laboratory safety parameters.
Change in concentration of BLZ-100 in the blood | Prior to dosing and at 10 minutes, 30 minutes, and 60 minutes post BLZ-100 administration
  BLZ-100 levels in blood will be analyzed by chemical means and these data will be used to calculate pharmacokinetic parameters.

SECONDARY OUTCOMES:
Fluorescence signal in excised central nervous system tumors | At least 1 hour post-dose
  Fluorescence signal in sections of excised tumor and adjacent normal tissue will be measured using an infrared imaging system.
Extent of resection (expansion cohort only) | At completion of surgery for surgeon assessment and up to 1 week after surgery for MRI assessment
  For subjects enrolled in the expansion cohort, an extent of resection assessment will be made by the surgeon and confirmed by post-operative MRI according to standard of care procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Leary, MD, MS, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's, Seattle, Washington, United States